CLINICAL TRIAL: NCT01944696
Title: Cycled Phototherapy: A Safer Effective Treatment for Small Premature Infants?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Stanford University (Other); Lucile Packard Children's Hospital (Other)
Responsible Party: Principal Investigator, Jon Edward Tyson, Professor, Vice Dean for Clinical Research and Healthcare Quality, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-13-0406
Record Dates: First submitted 2013-09-12; First posted 2013-09-18 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Hyperbilirubinemia; Premature Newborns; Extremely Low Birth Weight
Keywords: hyperbilirubinemia; prematurity; extremely low birth weight (ELBW); phototherapy; cycled phototherapy; intermittent phototherapy
MeSH Terms: conditions — Hyperbilirubinemia; Premature Birth | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- continuous (uninterrupted) phototherapy (Active Comparator): standard phototherapy
  Interventions: Other: phototherapy
- 15 minute per hour cycled phototherapy (Experimental): 15 minute per hour cycled phototherapy
  Interventions: Other: phototherapy

INTERVENTIONS:
Other: phototherapy — Cycled versus continuous phototherapy during the first 2 wks after birth, both administered at bilirubin thresholds used in the NICHD Neonatal Network Phototherapy trial .

SUMMARY:
Cycled (intermittent) phototherapy will be compared to continuous (uninterrupted) phototherapy in the treatment of hyperbilirubinemia (newborn jaundice) in extremely low birth weight newborns in a pilot randomized controlled trial.

Hypothesis: Cycled phototherapy (PT) will provide the same benefits as continuous phototherapy in extremely low birth weight (ELBW) infants without the risks that have been associated with continuous phototherapy.

DETAILED DESCRIPTION:
Phototherapy (PT) is widely used and assumed to be safe as well as effective in reducing total bilirubin (TB) levels. Our recent NICHD Network Trial showed that aggressive use of phototherapy reduces neurodevelopmental impairment (NDI), but may increase deaths among ELBW infants. Among ventilator treated infants <750 g birth weight (BW) (n =696), conservative Bayesian analyses (using a neutral prior probability) identified a 99% (posterior) probability that aggressive phototherapy reduced profound NDI but a 99% probability that it increased deaths relative to conservative phototherapy. The possibility that PT increases deaths among high risk infants is also suggested by the Collaborative Phototherapy trial (performed in the 1970s), the only large RCT in which LBW infants were randomly assigned to receive PT or no PT. The relative risk for death among those randomized to PT relative to those randomized to no PT was 1.32 (0.9-1.82) among all LBW infants and 1.49 (0.93-2.40) among ELBW infants. These findings are consistent with a major increase in mortality but have been ignored because the p was >0.05, an error often made in ignoring important potential treatment hazards when power is limited.

Multiple studies, most performed decades ago in larger infants, found that short on/off cycles of PT (e.g. 15 min on/60 min off, 1 h on/3 h off, or 1 h on/1 h off ) are as effective as uninterrupted PT to reduce TSB. (Cycles with >6 h off PT do not appear to be as effective as uninterrupted PT). The clinical use of uninterrupted rather than cycled PT appears to be based largely on the assumption that PT is safe for all infants.

ELIGIBILITY:
Inclusion Criteria:

* birth weight 401-1000 grams
* age less than or equal to 24 hours

Exclusion Criteria:

* hemolytic disease
* major anomaly
* overt nonbacterial infection

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Brain stem auditory evoked response wave V latency | 35 wks postmenstrual age or discharge
  a measure of transient or permanent bilirubin neurotoxicity

SECONDARY OUTCOMES:
Peak Total Serum Bilirubin (tsb) | 14 days from birth
  Total serum bilirubin (TSB) measurements will be obtained following a study protocol modeled on standard practice for monitoring TSB in ELBW newborns.

OTHER OUTCOMES:
Neurodevelopmental status | 2 years adjusted age
  The Network supports and assures carefully standardized neurodevelopmental testing at 2 years adjusted age for inborn ELBW patients. The reliability of these exams is verified annually in the Network. These assessments will provide data for survival rates without impairment
Survival | Before discharge from the neonatal ICU and at 2 years adjusted age
  The Neonatal Research Network supports and assures outcome assessment at 2 years adjusted age for inborn ELBW patients. These assessments will provide data for survival rates and survival rates without impairment

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Tyson, MD, Principal Investigator — The University of Texas Health Science Center, Houston; David K Stevenson, MD, Principal Investigator — Stanford School of Medicine
Locations (6):
- United States (6):
  - University of Alabama at Birmingham School of Medicine - UAB Hospital, Birmingham, Alabama
  - Stanford University - Lucile Packard Children's Hospital, Palo Alto, California
  - University of Cincinnati College of Medicine - Good Samaritan Hospital, Cincinnati, Ohio
  - The University of Texas Southwestern Medical School - Clements University Hospital, Dallas, Texas
  - The University of Texas Health Science Center at Houston; Memorial Hermann-TMC-NICU, Houston, Texas
  - The University of Texas Health Science Center at San Antonio - University Hospital, San Antonio, Texas

REFERENCES:
- [Background] Tyson JE, Pedroza C, Langer J, Green C, Morris B, Stevenson D, Van Meurs KP, Oh W, Phelps D, O'Shea M, McDavid GE, Grisby C, Higgins R; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Does aggressive phototherapy increase mortality while decreasing profound impairment among the smallest and sickest newborns? J Perinatol. 2012 Sep;32(9):677-84. doi: 10.1038/jp.2012.64. Epub 2012 May 31. PMID 22652561
- [Background] Hintz SR, Stevenson DK, Yao Q, Wong RJ, Das A, Van Meurs KP, Morris BH, Tyson JE, Oh W, Poole WK, Phelps DL, McDavid GE, Grisby C, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Is phototherapy exposure associated with better or worse outcomes in 501- to 1000-g-birth-weight infants? Acta Paediatr. 2011 Jul;100(7):960-5. doi: 10.1111/j.1651-2227.2011.02175.x. Epub 2011 Feb 25. PMID 21272067
- [Derived] Arnold C, Tyson JE, Pedroza C, Carlo WA, Stevenson DK, Wong R, Dempsey A, Khan A, Fonseca R, Wyckoff M, Moreira A, Lasky R. Cycled Phototherapy Dose-Finding Study for Extremely Low-Birth-Weight Infants: A Randomized Clinical Trial. JAMA Pediatr. 2020 Jul 1;174(7):649-656. doi: 10.1001/jamapediatrics.2020.0559. PMID 32338720